CLINICAL TRIAL: NCT03683953
Title: The Treatment of Bronchopulmonary Dysplasia by Intratracheal Instillation of Mesenchymal Stem Cells
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Women and Children Hospital (Other)
Responsible Party: Principal Investigator, yangjie, Professor, Guangdong Women and Children Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Guangdong W CH
Record Dates: First submitted 2018-09-24; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-07

CONDITIONS: Safety Issues; Effect of Drugs
Keywords: mesenchymal stem cells; safety; effect; BPD
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 0.9% sodium chloride intratracheal instillate on 14 days after birth
  Interventions: Drug: 0.9% sodium chloride
- mesenchymal stem cells (Experimental): mesenchymal stem cells intratracheal instillate on 14 days after birth ,dose is 25 million cells/kg
  Interventions: Other: mesenchymal stem cells therapy

INTERVENTIONS:
Other: mesenchymal stem cells therapy — mesenchymal stem cells treatement of BPD for safety and effect evaluation0.9% sodium chloride incontrol group
  Arms: mesenchymal stem cells
Drug: 0.9% sodium chloride — 0.9% sodium chloride in control group
  Arms: Placebo

SUMMARY:
To study the effect and saftey of intratracheal instillation of mesenchymal stem cells for treatment BPD

DETAILED DESCRIPTION:
This is a Phase 1 clinical trial that constitues two points cohorts with 100 participants per cohort who will receive instillation dose of mesenchymal stem cells-25 million cells/kg,with ventilation after 14 days.And the placebol will be 0.9% sodium choride. The investigator will proceed the groups during the same period.

1. Deographic Data and Baseline charateristics of the studied groups were collected:

   Gestational age (weeks) Birth weight (g) gender Cesarean section delivery Antenatal steroids Prolonged rupture of membrane Multiple pregnancies APGAR score at 5 minutes
2. mesenchymal stem cels dose is 25 million cells/kg
3. Assessment the incidence of BPD after instillation of Mesenchymal stem cells
4. the adverse after instillation of Mesenchymal stem cells

ELIGIBILITY:
Inclusion Criteria:

twenty-eight weeks to thirty-seven weeks prematures who need ventilaton for 14 days after birth, and the oxygen concentration is more than 30%

Exclusion Criteria:

Preterm infants with major congenital malformations, chromosomal anomalies, inborn errors of metabolism and clinical or laboratory evidence of a congenital infection

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2018-09-29 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
number of patients with BPD after instillation mesenchymal stem cells | up to 28 days after birth
  incidence of BPD

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yang, PHD, Principal Investigator — Guangzhou, Guangdong,China，511442

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mezey E, Nemeth K. Mesenchymal stem cells and infectious diseases: Smarter than drugs. Immunol Lett. 2015 Dec;168(2):208-14. doi: 10.1016/j.imlet.2015.05.020. Epub 2015 Jun 4. PMID 26051681